CLINICAL TRIAL: NCT03280368
Title: Adherence and the Role of Coagulation Assays in Patients Treated With Dabigatran Etexilate for Non-valvular Atrial Fibrillation
Brief Title: Adherence and Coagulation Assays in Dabigatran-treated Patients With Atrial Fibrillation
Acronym: ARCADE
Status: Completed | Type: Observational
Sponsor: Hospitalsenheden Vest (Other)
Collaborators: Catharina Ziekenhuis Eindhoven (Other); Siemens Corporation, Corporate Technology (Industry); Diagnostica Stago (Industry); Boehringer Ingelheim (Industry); European Society of Cardiology (Network); ANIARA (Unknown); University of Aarhus (Other); Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Willemijn Comuth, Cardiologist, PhD-fellow, Hospitalsenheden Vest
Other Study IDs: 1-16-02-191-14
Record Dates: First submitted 2016-10-26; First posted 2017-09-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Atrial Fibrillation; Medication Adherence; Blood Coagulation Tests; Anticoagulants; Circulating, Hemorrhagic Disorder; Drug Effect; Drug Use; Drug Toxicity; Drug Intolerance; Blood Clot; Blood Coagulation Disorder; Laboratory Problem; Bleeding; Thrombosis
MeSH Terms: conditions — Atrial Fibrillation; Medication Adherence; Hemorrhagic Disorders; Drug-Related Side Effects and Adverse Reactions; Thrombosis; Blood Coagulation Disorders; Hemorrhage | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- A healthy volunteers: Pre-clinical study. Healthy volunteers. Plasma pooled and spiked with dabigatran. Measurement of plasma concentration of dabigatran with liquid chromatography tandem mass-spectrometry and the anticoagulant effect of dabigatran using coagulation assays.
  Interventions: Other: Bloodtest
- A patients: Pre-clinical study. Patients with atrial fibrillation treated with dabigatran etexilate.
  Interventions: Other: Bloodtest
- B: Patients with an indication for treatment with dabigatran etexilate for atrial fibrillation and intended for electrocardioversion.
  Inclusion before initiation of anticoagulation.
  Interventions: Other: Bloodtest; Other: Questionnaires
- C: Patients with an indication for treatment with dabigatran etexilate for atrial fibrillation. Inclusion before initiation of anticoagulation.
  Interventions: Other: Bloodtest; Other: Questionnaires

INTERVENTIONS:
Other: Bloodtest
Other: Questionnaires
  Groups: B; C

SUMMARY:
In patients with non-valvular atrial fibrillation treated with dabigatran etexilate, the level of adherence will be measured using a questionnaire, the Danish National Prescription Registry and pillcount and will be related to plasma levels of dabigatran measured by liquid chromatography tandem mass spectrometry (LC-MS/MS) and coagulation assays. The aim of the study is to measure the level of adherence and evaluate the usefulness of different coagulation assays to measure adherence in these patients. Furthermore, the aim is to determine the correlation between the anticoagulant effect of dabigatran using different coagulation assays and plasma levels of dabigatran.

Most studies so far have been performed in vitro with plasma samples spiked with dabigatran. In this study the present knowledge from results of coagulation assays in dabigatran spiked plasma samples will be compared to the results of coagulation assays using blood samples from real-life patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Non-valvular atrial fibrillation
* Indication for dabigatran etexilate

Exclusion Criteria:

* Use of anticoagulant medication within the last month
* Contra-indication to dabigatran etexilate
* Unable or not wishing to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation with an indication for initiation of dabigatran etexilate
Sampling Method: Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2014-06; Primary Completion 2019-11 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Medication adherence Stability after storage at -80 degrees C; correlation between plasma concentration and the anticoagulant effect of dabigatran | 2 years
  Measured by pillcount, bloodtests, the Danish National Prescription Registry and the Morisky Medication Adherence Scale

SECONDARY OUTCOMES:
Patient treatment satisfaction | 2 years
  Measured by the Anticlot Treatment Scale
Medication persistence | 2 years
  Time from start to end of dabigatran treatment
Kidney function | 2 years
  Creatinine and Glomerular Filtration Rate calculated by the Cockroft Gault formula
Side-effects | 2 years
  Bleeding, gastrointestinal side-effects
Dabigatran plasma concentrations | 2 years
  Measured by liquid-chromatography tandem mass spectrometry (ng/mL)
Weight | 2 years
  kilograms
Height | 2 years
  meters
Waist circumference | 2 years
  centimeters
Prothrombin time | 2 years
  seconds
Activated partial thromboplastin time | 2 years
  seconds
ROTEM | 2 years
  Clotting time (seconds)
Diluted thrombin time (calibrated for dabigatran) | 2 years
  ng/mL
Ecarin chromogenic assay | 2 years
  ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Willemijn Comuth, MD, Principal Investigator — Hospitalsenheden Vest; Steen Husted, MD, PhD, Study Chair — Hospitalsenheden Vest
Locations (1):
- Hospital Unit West, Herning, Mid-Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Comuth WJ, de Maat MPM, van de Kerkhof D, Malczynski J, Husted S, Kristensen SD, Munster AB. Adherence to dabigatran etexilate in atrial fibrillation patients intended to undergo electrical cardioversion. Eur Heart J Cardiovasc Pharmacother. 2019 Apr 1;5(2):91-99. doi: 10.1093/ehjcvp/pvy047. PMID 30608563
- [Result] Comuth WJ, Lauridsen HH, Kristensen SD, Munster AB. Translation, Cultural Adaptation, and Psychometric Properties of the Danish Version of the Anti-Clot Treatment Scale. TH Open. 2018 Sep 13;2(3):e280-e290. doi: 10.1055/s-0038-1670631. eCollection 2018 Jul. PMID 31249952
- [Result] Comuth WJ, Henriksen LO, van de Kerkhof D, Husted SE, Kristensen SD, de Maat MPM, Munster AB. Comprehensive characteristics of the anticoagulant activity of dabigatran in relation to its plasma concentration. Thromb Res. 2018 Apr;164:32-39. doi: 10.1016/j.thromres.2018.02.141. Epub 2018 Feb 17. PMID 29475179